CLINICAL TRIAL: NCT00619281
Title: Prospective, Observational Study in Cardiac Surgery: How Much Cardiac Output is Enough?
Brief Title: How Much Cardiac Output is Enough?
Status: Completed | Type: Observational
Sponsor: Klinikum Ludwigshafen (Other)
Collaborators: Klinikum der Stadt Ludwigshafen, Department of Anesthesiology and Intensive Care Medicine (Unknown); Klinikum der Stadt Ludwigshafen, Department of Cardiac Surgery (Unknown)
Responsible Party: Andreas Lehmann, MD, Klilnikum der Stadt Ludwigshafen, Dept of Anesthesiology and Intensive Care Medicine
Other Study IDs: CI-11-2007; klilu-11-2007-alehmann
Record Dates: First submitted 2007-12-28; First posted 2008-02-20 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Low Cardiac Output Syndrome
Keywords: Cardiac surgery; Low cardiac output syndrome; Mortality; Morbidity
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oberservation: 600 consecutive patients undergoing cardiac surgery

SUMMARY:
Low output syndrome is a common complication in patients undergoing cardiac surgery. Its incidence was reported to be 2 to 6% [1]. Morbidity and mortality of low output syndrome is high and the costs for treating the disease are immense.

The primary objective of this prospective observational study is to define a threshold for a critically reduced cardiac output requiring immediate therapy.

DETAILED DESCRIPTION:
Low output syndrome is a common complication in patients undergoing cardiac surgery. Its incidence was reported to be 2 to 6% [1]. In patients suffering from low output syndrome cardiac output is severely reduced due to myocardial failure. Among other reasons for myocardial failure, ischemia, insufficient myocardial protection during aortic cross-clamping, and severely reduced ventricular function prior surgery are the most common risk factors for low output syndrome. Low output syndrome is treated with positive inotropic drugs and mechanical assist devices [2]. Morbidity and mortality of low output syndrome is high and the costs for treating the disease are immense.

If cardiac output cannot be increased cardiac failure persist and vital organs are hypoperfused. Critical and prolonged hypoperfusion results in single and multi organ failure. Until today a definite threshold for a critically reduced cardiac output or cardiac index requiring immediate therapy is not completely known. Cardiogenic shock is diagnosed by clinical signs and it is not diagnosed by cardiac output or cardiac index. The critical value for a severely reduces cardiac index was reported to be in a range of 1.75 to 2.5L/min/m² [3-5].

The primary objective of this prospective observational study in 600 patients undergoing cardiac surgery is to try to define a threshold for a critically reduced cardiac output or cardiac index requiring immediate therapy.

If cardiac output and cardiac index are not reduced below a critical threshold, morbidity, mortality, and length of stay in the intensive care unit and in the hospital are reduced [6].

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery,
* Written informed consent

Exclusion Criteria:

* Missing consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 600 patients undergoing cardiac surgery
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to try to define a threshold value for a critically reduced cardiac output or cardiac index requiring immediate therapy to reduce mortality and morbidity. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Boldt, MD, Study Director — Klinikum Ludwigshafen, Department of Anesthesiology and Intensive Care medicine
Locations (1):
- Klinikum der Stadt Ludwigshafen, Department of Anesthesiology and Intensive Care Medicine, Ludwigshafen, Germany

REFERENCES:
- [Background] Hausmann H, Potapov EV, Koster A, Krabatsch T, Stein J, Yeter R, Kukucka M, Sodian R, Kuppe H, Hetzer R. Prognosis after the implantation of an intra-aortic balloon pump in cardiac surgery calculated with a new score. Circulation. 2002 Sep 24;106(12 Suppl 1):I203-6. PMID 12354734
- [Background] Lehmann A, Boldt J. New pharmacologic approaches for the perioperative treatment of ischemic cardiogenic shock. J Cardiothorac Vasc Anesth. 2005 Feb;19(1):97-108. doi: 10.1053/j.jvca.2004.11.020. No abstract available. PMID 15747280
- [Background] Bohrer H, Schmidt H, Motsch J, Gust R, Bach A, Martin E. Gastric intramucosal pH: a predictor of survival in cardiac surgery patients with low cardiac output? J Cardiothorac Vasc Anesth. 1997 Apr;11(2):184-6. doi: 10.1016/s1053-0770(97)90211-1. PMID 9105990
- [Background] Hochman JS, Sleeper LA, Webb JG, Sanborn TA, White HD, Talley JD, Buller CE, Jacobs AK, Slater JN, Col J, McKinlay SM, LeJemtel TH. Early revascularization in acute myocardial infarction complicated by cardiogenic shock. SHOCK Investigators. Should We Emergently Revascularize Occluded Coronaries for Cardiogenic Shock. N Engl J Med. 1999 Aug 26;341(9):625-34. doi: 10.1056/NEJM199908263410901. PMID 10460813
- [Background] Adams HA, Baumann G, Gansslen A, Janssens U, Knoefel W, Koch T, Marx G, Muller-Werdan U, Pape HC, Prange W, Roesner D, Standl T, Teske W, Werner G, Zander R; I.A.G.-Schock. [Definition of shock types]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2001 Nov;36 Suppl 2:S140-3. doi: 10.1055/s-2001-18174. German. PMID 11753724
- [Background] Polonen P, Ruokonen E, Hippelainen M, Poyhonen M, Takala J. A prospective, randomized study of goal-oriented hemodynamic therapy in cardiac surgical patients. Anesth Analg. 2000 May;90(5):1052-9. doi: 10.1097/00000539-200005000-00010. PMID 10781452